CLINICAL TRIAL: NCT05540496
Title: Ocular, Periocular and Cutaneous Tolerance and Efficacy of Formula 2039002 10 Product in Patients With Palpebral Eczema During 4 Weeks Under Dermatological and Ophthalmological Controls
Brief Title: Ocular, Periocular and Cutaneous Tolerance and Efficacy of Formula 2039002 10 in Patients With Palpebral Eczema
Status: Completed | Type: Observational
Sponsor: Cosmetique Active International (Industry)
Responsible Party: Sponsor
Other Study IDs: LRP20015-TOLERIANE ULTRA YEUX
Record Dates: First submitted 2022-09-08; First posted 2022-09-14 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-09

CONDITIONS: Eczema Eyelid
Keywords: palpebral eczema; ocular; periocular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The eyelids are particularly susceptible to eczema. Eyelid eczemas also called palpebral eczema, are a common condition that causes the skin on or around the eyelid to become dry, itchy, and irritated.

The study aims at evaluating the ocular and peri-ocular tolerance and the efficacy of the investigational product under normal conditions of use in participants with a palpebral eczema ground.

This open-labeled, multicentric study was conducted under dermatological and ophthalmological control in Caucasian subjects over 18 years of age, of all skin types and having a sensitive skin, especially on eye contour. The investigational product was to be applied twice daily on eyes contour for 4 weeks.

DETAILED DESCRIPTION:
The evaluation of the investigational product in participants with a palpebral eczema ground has been conducted under dermatological and ophthalmological control by Dermatech.

The study was conducted in the spirit of the French and European Guidelines for Good Clinical Practice, the recommendations of the International Conference on Harmonization (ICH) and according to the Helsinki Declaration in its latest version (Seoul 2008) and the General Data Protection Regulation (GDPR).

A 35-patient panel is considered as enough size to reach study objectives. The following statistical analysis are performed after data control and randomisation released.

* Excluded data: In case of incoherent /aberrant value, it could be decided to exclude the data from the analysis (a justification will be brought).
* Protocol deviation: All deviations from the protocol are listed. Deviations that may have an impact on the study results are identified.
* Initial characteristics: The initial characteristics of the patients will be summarized using descriptive statistics (means, minimum and maximum values for quantitative variables, absolute and relative frequencies for qualitative variables).
* Clinical assessment and self-assessment scales:

  * Calculation of mean and standard deviation at each time point at Day0 Time0 (D0T0), Day0 Time10 minutes (D0T10min), D14 and Day28 Time0 (D28T0) for the clinical assessment and at D0T0, D14 and D28T0 for the self-assessment scales.
  * Evaluation of time effect using a linear mixed effect model, with time (at D0T0, D0T10min, D14 and D28T0 for the clinical assessment and at D0T0, D14 and D28T0 for the self-assessment scales) as a fixed effect, and patients as a random effect to take into account that several measurements were performed on each patient.
  * In case of significance of the time effect, multiple comparisons among timepoints will be performed with Tukey adjustment). In case of non-convergence of the linear mixed effect model, a logistic mixed effect model could be performed as an alternative, where modalities would be grouped into two modalities (presence/absence of sign).
* Questionnaire of cosmetic acceptability: Calculation of effective and percentages of positive answers.
* Quality of life questionnaires: Qualitative variables will be summarized by effective and percentages. Quantitative variables will be summarized by mean and standard deviation, median and quartiles, and range.
* Safety analysis: Interpretation of safety data was performed by analyzing each reaction, attributable to the application of study product (reactions reported by patient in the daily log questionnaire and reactions reported by investigator during examination). The investigator gives his conclusion on the investigational product cutaneous acceptability.

Regarding the participants, the reasons for which a participant can be discontinued from the study or withdrawn from the data analysis, are:

* Withdrawal of the participant's consent (possible at any time and for whatever reason): in this case, the data collected for the study up to the date of the withdrawal will be analyzed unless patient express opposition. Patient agreement will be sought by the investigator or the study responsible for the use of routine follow-up data that could be collected after withdrawal of consent.
* Lost to follow up: in this case, the investigator or the study responsible will make an effort to contact the participant and determine the reason (at least 2 calls reported in the Case Report Form (CRF)).
* Emergence of a non-inclusion criterion.
* Investigator or study responsible decision (for example but not limited to: the investigator or study responsible believes for safety reasons or in the best interest of the participant that he/she had to stop its study participating).
* Protocol violation. The reason(s) of participant premature release will be sought and documented by the investigator or the study responsible in the appropriate pages of the CRF.

Regarding the investigational product, expected reactions after application of this type of cosmetic product are slight to very slight and not persistent discomfort or irritation reaction and are not considered as adverse events (AE). All adverse events will be investigated and evaluated from the informed consent form signature date for the study last visit date.

If such an adverse event is on-going at the final visit, the investigator will follow the event until complete resolution or stabilization.

ELIGIBILITY:
Inclusion Criteria:

* caucasian
* phototype I to IV
* palpebral eczema ground (blepharitis, epiphora, chronic whimpering/watery eyes)
* sensitive skin and especially on eye contour
* all skin types of eyes contours
* not tanned on the face (no sun or artificial U.V. exposure for at least a month)
* no exfoliation, scrubbing or peeling of the whole face for at least 2 weeks

Exclusion Criteria:

* at least one ocular functional sign at inclusion day
* receiving a medication which, in the investigator's judgment, places the patient at undue risk
* an intra-ocular surgery within the 6 months preceding the beginning of the study
* an ocular laser session, within the month preceding the beginning of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: participants with palpebral eczema meeting the inclusion and exclusion criteria and agreeing with the study constraints
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2021-04-17 (Actual); Study Completion 2021-04-17 (Actual)

PRIMARY OUTCOMES:
change in clinical assessment of efficacy items | change from baseline to Day28 Time0
  irritated aspect of the eye contours, swelling of eye contours on a 6-point scale

SECONDARY OUTCOMES:
change in dermatological evaluation of the tolerance - functional signs | change from baseline to Day28 Time10minutes
  collection of functional signs of peri-ocular area skin (by asking the patient): prickling, tightness, itching, sensations of heat/burn on a 6-point scale
change in dermatological evaluation of the tolerance - clinical signs | change from baseline to Day28 Time10minutes
  examination of clinical signs of peri-ocular area (observed by the dermatologist): erythema, edema, desquamation/dryness, roughness, eczematide, palpebral swelling on upper and lower eyelid, others (papules, blisters of skin) on a 6-point scale
change in ophthalmological evaluation of the tolerance - functional signs | change from baseline to Day28 Time10minutes
  functional signs performed on a 6-point scale on the eyes and the lid margin
change in ophthalmological evaluation of the tolerance - physical signs | change from baseline to Day28 Time10minutes
  Examination of the lid margin, the bulbar conjunctiva, the tarsal conjunctiva, the cornea and the tear film
change in self-assessment of efficacy items | change from baseline to Day28 Time0
  soothing feeling of eye contours, swelling feeling of eye contours, irritated aspect of eye contours on a 6-point scale (0= none to 5= very high)
change in quality of life | change from baseline to Day28 Time0
  Dermatology Life Quality Index (DLQI) questionnaire covering 6 domains: symptoms and feelings, daily activities, leisure, work and school, personal relationships, and treatment
change in sensitivity and quality of life of patients | change from baseline to Day28 Time0
  occurrences during the previous week (like presence of eye contour redness, presence of eye contour discomfort ...), quality of life deterioration, factors inducing cutaneous sensitivity (like sun exposure, wind exposure...)
cutaneous acceptability and efficacy | Day28 Time0
  18 questions using the scale "Agree", "Quite agree", "Quite disagree", "Disagree" or "No opinion"
global acceptability of the ocular and peri-ocular area | Day28
  evaluation of the global acceptability of the ocular and peri-ocular area by the ophthalmologist and dermatologist using the following scale : very good (no reaction), good (expected manifestations of this type of product), moderate (not expected manifestations for a few patients), bad (not expected manifestations for the majority of patients)

CONTACTS AND LOCATIONS:
Overall Officials: Meryem Nili, Study Director — Dermatech
Locations (2):
- Georgia (2):
  - LTD Health, Batumi
  - LTD Kutaisi Primary Health Care centre #1, Kutaisi

REFERENCES:
- [Derived] Tan J, Demessant A, Le Dantec G, Le Floc'h C, Kerob D. Tolerance and Efficacy of a Dermocosmetic Containing Neurosensine(R) in Subjects with Eyelid Eczema. Clin Cosmet Investig Dermatol. 2023 Jan 20;16:161-165. doi: 10.2147/CCID.S391890. eCollection 2023. PMID 36711070